CLINICAL TRIAL: NCT00720057
Title: A Multicenter, Double-Blind, Randomized, Parallel, Placebo-Controlled Trial Assessing the Analgesic Efficacy of a Single, Oral Dose of an Extended Release Naproxen Sodium Tablet in Postsurgical Dental Pain
Brief Title: Assessing the Analgesic Efficacy of Naproxen Sodium in Postsurgical Dental Pain.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13130; 2014-005269-66 (EudraCT Number)
Record Dates: First submitted 2008-07-01; First posted 2008-07-22 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Toothache
Keywords: Dental Pain; Analgesia
MeSH Terms: conditions — Toothache; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naproxen sodium ER (BAYH6689) (Experimental): single dose (1 tablet) ER Naproxen sodium 660 mg with a full glass of water (240ml) within 1 - 4 hours post dental surgery.
  Interventions: Drug: Naproxen Sodium ER (BAYH6689)
- Placebo (Placebo Comparator): Single dose (1 tablet) of placebo with a full glass of water (240ml) within 1 - 4 hours post dental surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen Sodium ER (BAYH6689) — Analgesic efficacy in dental pain; per oral; 1 tablet extended release Naproxen Sodium; with a full glass of water within 4 hours post surgery
  Arms: Naproxen sodium ER (BAYH6689)
Drug: Placebo — Inactive ingredient; per oral; 1 lactose based tablet; with a full glass of water within 4 hours post surgery
  Arms: Placebo

SUMMARY:
To evaluate the analgesic efficacy of a single, oral dose of a naproxen sodium extended-release tablet, compared to placebo in postsurgical dental pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male and female volunteers between 16 to 45
* Scheduled to undergo surgical removal of 1 - 2 impacted third molars, one of which must be at least a partial mandibular bony impaction
* No use of any analgesics, nonsteroidal anti-inflammatory drugs (NSAIDs), aspirin, any other pain reliever (Over The Counter or prescription), or herbal supplements within 5 days of surgery
* Have moderate to severe postoperative pain on the Categorical Pain Intensity Scale (a score of at least 2 on a 4 point scale) and a score of >/= 50 mm on the 100-mm visual analog Pain Severity Rating Scale

Exclusion Criteria:

* History of hypersensitivity to naproxen sodium, aspirin (ASA), other NSAIDs, opioid analgesics, and similar pharmacological agents or components of the investigational products, including the placebo
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases, or malignancies
* Relevant concomitant disease such as asthma (exercise induced asthma is permitted), chronic sinusitis or nasal structural abnormalities causing greater than 50 percent obstruction (polyposis nasi, marked septal deviation) that can interfere with the conduct of the study
* Current or past history of bleeding disorder(s)
* History of gastrointestinal bleeding or perforation, related to previous NSAID therapy. Active, or history of recurrent peptic ulcer/hemorrhage (two or more distinct episodes of proven ulceration or bleeding)

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 312 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Austin, Texas
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Laurora I, An R. Efficacy of single-dose, extended-release naproxen sodium 660 mg in postsurgical dental pain: two double-blind, randomized, placebo-controlled trials. Curr Med Res Opin. 2016;32(2):331-42. doi: 10.1185/03007995.2015.1123680. Epub 2015 Dec 15. PMID 26588111
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Screening Period occurred up to 28 days prior to the day of dental surgery. A total of 447 subjects were screened, of which 135 were excluded (72 did not meet inclusion criteria, 19 refused to participate, 44 other reasons); 312 subjects were randomized and included in the intent-to-treat (ITT) population for efficacy and safety analysis.
Period: Overall Study
Arm/Group | Naproxen Sodium ER (BAYH6689) | Placebo
Started | 153 | 159
Completed | 152 | 156
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Sodium ER (BAYH6689) | Placebo | Total
Number analyzed (Participants) | 153 | 159 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.8 (4.03) | 20.4 (4.31) | 20.6 (4.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 106 | 195
  Male | 64 | 53 | 117
Baseline Pain Intensity by Categorical Scale [Number; unit: participants] — Categorical scale: No Pain (0), Mild Pain (1), Moderate Pain (2), Severe Pain (3).
  participants
    Moderate | 99 | 103 | 202
    Severe | 54 | 56 | 110
Baseline Pain Intensity by Visual Analog Scale [Mean (Standard Deviation); unit: scores on a scale] — Visual Analog Scale 0-100 mm: 0 is no pain and 100 is worse possible pain.
  scores on a scale | 72.3 (13.13) | 72.6 (11.91) | 72.4 (12.51)

OUTCOME MEASURES:

1. Primary Outcome: Summed Pain Intensity Difference (SPID)
Description: Categorical pain intensity scale - no pain (0), mild pain (1), moderate pain (2), or severe pain (3) was used for all pain intensity assessments postdose. Time-weighted Sum Pain Intensity Difference (SPID) was calculated by multiplying the Pain Intensity Difference (PID) score at each postdose time point by the duration (in hours) since the preceding time point and then summing these values over 0-24 and 16-24 hours, respectively.
Time Frame: 0 to 24 hours post dose
Population: Randomized population is defined as all subjects who signed informed consent form, completed the screening period, and were randomized. The ITT population is defined as all subjects who were randomized and received at least one dose of the study treatment. Efficacy analyses are based on the ITT population (n=312).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naproxen Sodium ER (BAYH6689) | Placebo
Number analyzed (Participants) | 153 | 159
units on a scale
  SPID 0-24 | 25.9 (25.87) | -3.1 (18.40)
  SPID16-24 | 8.8 (9.30) | -1.0 (6.89)
Statistical Analysis 1: Comparison: Naproxen Sodium ER (BAYH6689) vs Placebo; The treatment differences between the two groups were tested each at the 5% two-sided significant level using a hierarchal testing procedure to control the overall type 1 error. SPID16-24 was eligible for testing only after a statistically significant difference between the two arms with respect to SPID0-24 was observed. The SPIDs were analyzed via ANCOVA model with treatment and trial site as fixed effects and baseline pain intensity score as the covariate; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Secondary Outcome: Total Pain Relief (TOTPAR)
Description: Pain relief categorical rating scale - no relief (0), a little relief (1), some relief (2), a lot of relief (3), or complete relief (4) was used for all pain relief assessments postdose. Time weighted total pain relief (TOTPAR) was calculated by multiplying the pain relief score at each postdose time point by the duration (in hours) since the preceding time point and then summing these values.
Time Frame: 0-24 hours post dose
Population: Efficacy analyses were based on ITT population (n=312).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naproxen Sodium ER (BAYH6689) | Placebo
Number analyzed (Participants) | 153 | 159
units on a scale
  TOTPAR 0 - 6 hours | 12.7 (7.81) | 3.1 (5.07)
  TOTPAR 0 - 12 hours | 25.5 (17.06) | 5.5 (10.70)
  TOTPAR 0 - 16 hours | 34.1 (23.49) | 7.2 (14.83)
  TOTPAR 0 - 24 hours | 51.3 (36.41) | 10.9 (23.95)
  TOTPAR 16 - 24 hours | 17.2 (13.37) | 3.7 (9.40)
Statistical Analysis 1: Comparison: Naproxen Sodium ER (BAYH6689) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

3. Secondary Outcome: Summed Pain Intensity Difference at Specific Time Intervals
Description: Categorical pain intensity scale - no pain (0), mild pain (1), moderate pain (2), or severe pain (3) was used for all pain intensity assessments postdose. Time-weighted Sum Pain Intensity Difference (SPID) was calculated by multiplying the Pain Intensity Difference (PID) score at each postdose time point by the duration (in hours) since the preceding time point and then summing these values for 0-6, 0-12, 0-16 hour intervals, respectively.
Time Frame: 0-16 hours post dose
Population: Efficacy analyses were based on ITT population (n=312).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naproxen Sodium ER (BAYH6689) | Placebo
Number analyzed (Participants) | 153 | 159
units on a scale
  SPID 0 - 6 | 6.2 (5.7) | -0.4 (4.2)
  SIPD 0 - 12 | 12.7 (12.3) | -1.4 (8.54)
  SIPD 0 - 16 | 17.1 (16.85) | -2.0 (11.68)
Statistical Analysis 1: Comparison: Naproxen Sodium ER (BAYH6689) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

4. Secondary Outcome: Time to First Use of Rescue Medication
Description: Time to first use of rescue medication was estimated using the Kaplan-Meier method and analyzed by a Log rank test stratified by trial site and baseline pain intensity (PI). The outcome measure is time to first use of rescue medication. The criteria are if adequate pain relief is not achieved, then subjects are permitted to take rescue medication.
Time Frame: postdose to first use of rescue medication
Population: Efficacy analyses are based on ITT population (n=312).
Measure: Median (Full Range); unit: hours
Arm/Group | Naproxen Sodium ER (BAYH6689) | Placebo
Number analyzed (Participants) | 153 | 159
hours | 22.27 [1.07 to 22.27] | 1.90 [1.03 to 10.12]
Statistical Analysis 1: Comparison: Naproxen Sodium ER (BAYH6689) vs Placebo; The statistics are from the Kaplan-Meier method. The median for naproxen treatment arm was not estimable from Kaplan-Meier method, therefore it is presented as the maximum value from the full range; Test type: Superiority or Other; p < 0.001, Log Rank

5. Secondary Outcome: Global Assessment of the Investigational Product as a Pain Reliever
Description: Categorical Scale: Poor (0), Fair (1), Good (2), Very Good (3), Excellent (4).
Time Frame: at 24 hours postdose or immediately before first use of rescue medication
Population: Efficacy analyses are based on ITT population (n=312).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naproxen Sodium ER (BAYH6689) | Placebo
Number analyzed (Participants) | 153 | 159
units on a scale | 2.3 (1.43) | 0.6 (1.04)
Statistical Analysis 1: Comparison: Naproxen Sodium ER (BAYH6689) vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

6. Secondary Outcome: Time to Onset of Effect
Description: Time to onset of effect is defined as the time to meaningful pain relief, provided that the subjects experienced both "perceptible" and "meaningful" pain relief. Perceptible pain relief was defined as when the subject first began to feel any pain-relieving effect from the investigational product. Meaningful pain relief was defined as when the subject felt the degree of pain relief was meaningful to them.
Time Frame: from postdose to onset of first perceptible and meaningful pain relief for up to 6 hours
Population: Efficacy analyses are based on ITT population (n=312).
Measure: Median (Full Range); unit: hours
Arm/Group | Naproxen Sodium ER (BAYH6689) | Placebo
Number analyzed (Participants) | 153 | 159
hours | 1.37 [0.07 to 4.98] | 4.13 [0.07 to 4.75]
Statistical Analysis 1: Comparison: Naproxen Sodium ER (BAYH6689) vs Placebo; Test type: Superiority or Other; p < 0.001, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the treatment period through 5 days after investigational product or placebo administration. All Serious Adverse Events were collected through about 30 days after the last dose of investigational product or placebo.
Arm/Group | Naproxen Sodium ER (BAYH6689) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/153 | 0/159
Other Adverse Events (participants affected / at risk) | 10/153 | 36/159
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium ER (BAYH6689) (N=153) | Placebo (N=159)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (2)
Eye Swelling (Eye disorders) | 1 (1) | 0 (0)
Scotoma (Eye disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 24 (24)
Stomach Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth Socket Haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 14 (14)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Abscess Oral (Infections and infestations) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 8 (8)
Headache (Nervous system disorders) | 5 (5) | 6 (6)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less